CLINICAL TRIAL: NCT07335159
Title: Does Patient Testimonial Improve the Pain Relief Derived From a Brief Behavioral Intervention Delivered to Patients Experiencing Pain in a Clinic Waiting Room
Brief Title: Does Patient Testimonial Improve the Pain Relief Derived From a Brief Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004916_Testimonial
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pain; Acute Pain; Chronic Pain; Pain Management
MeSH Terms: conditions — Pain; Acute Pain; Chronic Pain; Agnosia | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Psychoeducation (Active Comparator): In the pain psychoeducation intervention, participants will be randomized to listen to a four-minute recording about different pain management strategies (e.g., ice, rest) to promote overall well-being.
  Interventions: Behavioral: Pain Psychoeducation
- Mindfulness (Experimental): In the mindfulness intervention, participants will be randomized to listen to 1 minute of psychoeducation about mindfulness that includes a patient testimonial, 1 minute of mindful breathing, 1 minute of mindful mapping (i.e., mindfulness of pain), and 1 minute of mindfulness of personal meaning.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Pain Psychoeducation — In the pain psychoeducation intervention, participants will be randomized to listen to a four-minute recording about different pain management strategies (e.g., ice, rest) to promote overall well-being.
  Arms: Pain Psychoeducation
Behavioral: Mindfulness — In the mindfulness intervention, participants will be randomized to listen to 1 minute of psychoeducation about mindfulness that includes a patient testimonial, 1 minute of mindful breathing, 1 minute of mindful mapping (i.e., mindfulness of pain), and 1 minute of mindfulness of personal meaning.
  Arms: Mindfulness

SUMMARY:
This project is a single-site, two-arm, randomized controlled trial investigating whether providing patients in an orthopedic clinic waiting room an audio-recorded mindfulness practice decreases their pain relative to an injury management control condition.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment at Tallahassee Orthopedic Center
* Understanding English instructions fluently
* Being 18 years of age or older

Exclusion Criteria:

* Unable to consent because of physical or mental incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Change in acute pain unpleasantness will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain unpleasantness.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Change in acute pain intensity will be measured with an individual item ("How much pain do you have, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain intensity.

OTHER OUTCOMES:
Interest in additional pain management resources | Immediately after the 4-minute audio recording
  After the recording, participants will complete a single dichotomous (yes/no) item assessing interest in additional pain management resources: "Would you like access to additional pain management resources similar to the one presented today?"
Net Promoter Scale | Immediately after the 4-minute audio recording
  The Net Promoter Scale (NPS) is a single-item measure of satisfaction and loyalty that asks respondents to rate how likely they are to recommend a product, service, or experience to others, typically on an 11-point scale from 0 ("not at all likely") to 10 ("extremely likely"). Responses are categorized as detractors (0-6), passives (7-8), or promoters (9-10). The overall NPS score is calculated by subtracting the percentage of detractors from the percentage of promoters, yielding a score ranging from -100 to +100.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No